CLINICAL TRIAL: NCT05797116
Title: Preoperative Multidisciplinary Team Meetings for High Risk Noncardiac Surgical Patients: A Nationwide Survey on Practice Variation, Facilitators and Barriers
Brief Title: Practice Variation in Preoperative MDT Meetings
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-16058
Record Dates: First submitted 2023-02-01; First posted 2023-04-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Multidisciplinary Communication; Preoperative Care; Patient Care Team
Keywords: multidisciplinary team meeting; high risk surgical patients; preoperative
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anaesthesiologists in the Netherlands: The participants in this study are anesthesiologists in the Netherlands, preferably those in charge of preoperative screening. One anesthesiologist per anesthesiology department may be included.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — 29-item Dutch survey about the implementation and practice variation of preoperative multidisciplinary team (MDT) meetings for high risk noncardiac surgical patients in the Netherlands.

SUMMARY:
The goal of this observational survey study is to evaluate the current practice variations of preoperative multidisciplinary team meetings (MDT meetings) for high risk noncardiac surgical patients. The main questions it aims to answer are:

* What is the current variation in Dutch hospitals in the practice of preoperative MDT meetings for high risk noncardiac surgical patients?
* Which facilitators and barriers influence the implementation process of preoperative MDT meetings? Participants are anesthesiologists in Dutch hospitals who will be asked to fill in a one-time survey. One anesthesiologist per anesthesiology department will be asked to fill in the survey. The survey will take approximately 5 to 10 minutes to complete.

DETAILED DESCRIPTION:
The number of patients with multiple comorbidities is significantly growing. Medical advances have made it possible to perform challenging surgical interventions to increase life expectancy. Yet, it is this group of patients that has a high risk of complications after a surgical intervention leading to a reduction in their quality of life and self-sustainability. Current European and Dutch guidelines recommend the implementation of preoperative multidisciplinary team (MDT) meetings for high risk noncardiac surgical patients. However, the evidence underlying the guideline recommendations is scarce. Furthermore, the implementation process of a well-functioning MDT meeting can be a challenge and may sometimes lead to no MDT meeting at all. And finally, the guidelines do not specify conditions by who or how the MDT meeting should be done, for example required attending specialties or specific subjects to be discussed. A broad practice variation in preoperative MDT meetings might thus be present and could be a complicating factor in the equal treatment of patients compliant to 'best practice'. The current survey will evaluate practice variation of preoperative MDT meetings for high risk noncardiac surgical patients in the Netherlands and assess possible facilitators and barriers in the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as anesthesiologist in a Dutch hospital

Exclusion Criteria:

* No informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The participants in this study are anesthesiologists in the Netherlands, preferably those in charge of preoperative screening. One anesthesiologist per anesthesiology department may be included.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of anaesthesia departments who employ preoperative multidisciplinary team (MDT) meetings for high risk noncardiac surgical patients in Dutch hospitals. | Baseline
  Percentage of anaesthesia departments who employ preoperative multidisciplinary team (MDT) meetings in which an anaesthesiologist is present, for high risk noncardiac surgical patients in Dutch hospitals.

SECONDARY OUTCOMES:
Frequency of multidisciplinary team (MDT) meetings per month | Baseline
  An approximate frequency of preoperative multidisciplinary team (MDT) meetings for high risk noncardiac surgical patients per month
Number of patients discussed per multidisciplinary team (MDT) meeting | Baseline
  Number of patients discussed per multidisciplinary team (MDT) meeting (average)
Duration of multidisciplinary team (MDT) meeting in minutes | baseline
  Duration of multidisciplinary team (MDT) meeting in minutes (average)

CONTACTS AND LOCATIONS:
Overall Officials: Carine JM Doggen, PhD, Principal Investigator — Rijnstate Hospital; Benedikt Preckel, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Rijnstate Hospital, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made accessible on request after agreement has been received from the entire project group. The principal investigator will communicate data availability with researchers sending the requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 12 months after publication
Access Criteria: Data will be made accessible on request after agreement has been received from the entire project group.